CLINICAL TRIAL: NCT01939639
Title: The Influence of Oxytocin on the Processing of Social Contact
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University Hospital, Bonn (Other)
Responsible Party: Principal Investigator, Rene Hurlemann, MD PhD M.Sc., University Hospital, Bonn
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: OXT_PS_2013; PS_2013 (Other Grant/Funding Number: University of Bonn)
Record Dates: First submitted 2013-08-27; First posted 2013-09-11 (Estimated); Last update posted 2013-09-11 (Estimated); Status verified 2013-09

CONDITIONS: Healthy Male Volunteers
Keywords: Oxytocin; fMRI
MeSH Terms: interventions — Oxytocin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Oxytocin (Experimental): 24 IU Oxytocin, intranasal application 30 min prior to the experiment
  Interventions: Drug: Oxytocin
- Placebo (Placebo Comparator): intranasal application, sodium chloride solution, 3 puffs per nostril
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Placebo — intranasal application, sodium chloride solution, 3 puffs per nostril
  Arms: Placebo
Drug: Oxytocin — 24 IU Oxytocin, intranasal application 45 min prior to the experiment
  Other Names: Syntocinon
  Arms: Oxytocin

SUMMARY:
Social touch can convey the most potent and salient of socio-emotional signals. While the hypothalamic peptide oxytocin (OXT) has been identified as a key neurochemical mediator of grooming in some other social species, its modulatory influence on human interpersonal touch is unknown. The investigators expect that OXT augments the hedonic value of touch and that this behavioral effect is paralleled at the neural level by an increased response in brain areas mediating rewarding aspects of social touch.

ELIGIBILITY:
Inclusion Criteria:

Healthy male volunteers

Exclusion Criteria:

Current or past psychiatric disease Current or past physical illness Psychoactive medication Tobacco smokers

Ages: 18 Years to 60 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2013-03; Primary Completion 2013-06 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
Pleasantness ratings of social touch | 30 minutes after the nasal spray administration
  After each trial, subjects are asked to use a visual analog scale to rate the pleasantness of the administered touch.
Blood-oxygen-level dependent signal in response to social touch | 30 minutes after the nasal spray administration
  By using functional magnetic resonance imaging we want to examine oxytocin's effects on the neural correlates (BOLD signal) of social touch.

SECONDARY OUTCOMES:
Questionnaire measurement of mood (PANAS) and anxiety (STAI). | 15 minutes before the nasal spray administration and (on average) 10 minutes after the fMRI experiment

OTHER OUTCOMES:
Saliva oxytocin concentrations | 15 minutes before the nasal spray administration and (on average) 10 minutes after the fMRI experiment

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Psychiatry, University of Bonn, Bonn, North Rhine-Westphalia, Germany

REFERENCES:
- See also: Related Info — http://renehurlemann.squarespace.com/welcome/